CLINICAL TRIAL: NCT01182116
Title: A Randomized, Controlled Trial to Compare the Functional Outcome and Quality of Life in Patients With Low Rectal Cancer Who Undergo a J Pouch or a Side to End Coloanal Anastomosis
Brief Title: Quality of Life in Patients That Undergo J Pouch or Side to End Coloanal Anastomosis for Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Massarat Zutshi, MD, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 08-178
Record Dates: First submitted 2010-05-25; First posted 2010-08-16 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Rectal Cancer
Keywords: J pouch; colorectal; rectal cancer; coloplasty
MeSH Terms: conditions — Rectal Neoplasms | interventions — Colonic Pouches

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- J Pouch side to end (Experimental): Colorectal surgery Function Quality of Life
  Interventions: Procedure: J Pouch

INTERVENTIONS:
Procedure: J Pouch — Comparing J pouch, side to end coloanal surgery

SUMMARY:
The investigators hypothesis is that the patients who receive a side to end anastomosis have bowel outcome and quality of life that is equivalent to those who receive a J pouch.

DETAILED DESCRIPTION:
The side to end anastomosis has become popular in recent years as it is technically simple to construct. The difference between the Baker type(side to end) of anastomosis and the J pouch, is that no formal pouch is constructed in the side to end. It has one staple line and the anastomosis.

The investigators hypothesis is that the patients who receive a side to end anastomosis have bowel outcome and quality of life that is equivalent to those who receive a J pouch.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with distal rectal cancers who will be having an abdominal proctocolectomy with a low colorectal anastomosis within 4 cm of the dentate line or a coloanal anastomosis will be candidates for this study.
2. No evidence of distant metastatsis -

Exclusion Criteria: Stage IV rectal cancer

1. History of radiation to the pelvis ( eg. for uterine or prostatic cancer)
2. Evidence of synchronus or metachronus disease
3. H/o dementia
4. Prisoners
5. Women who are pregnant
6. History of previous Right Colectomy
7. History of inflammatory bowel disease -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Improved function and capacity of the neorectum. | 2 years from date of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Massarat Zutshi, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parc Y, Ruppert R, Fuerst A, Golcher H, Zutshi M, Hull T, Tiret E, Hemminger F, Galandiuk S, Fender S, Weber K, Zimmerman A, Aiello A, Fazio V. Better Function With a Colonic J-Pouch or a Side-to-end Anastomosis?: A Randomized Controlled Trial to Compare the Complications, Functional Outcome, and Quality of Life in Patients With Low Rectal Cancer After a J-Pouch or a Side-to-end Anastomosis. Ann Surg. 2019 May;269(5):815-826. doi: 10.1097/SLA.0000000000003249. PMID 30921049